CLINICAL TRIAL: NCT05857098
Title: Detection of Local Field Potentials in the Ventral Tegmental Area of the Midbrain in Chronic Cluster Headache Patients Treated by Deep Brain Stimulation : a Feasibility Study
Brief Title: Detection of Local Field Potentials in the Ventral Tegmental Area of the Midbrain in Chronic Cluster Headache Patients
Acronym: DETECT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM23_0056
Record Dates: First submitted 2023-04-05; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-04

CONDITIONS: Cluster Headache; Trigeminal Autonomic Cephalgia
Keywords: Hypothalamus; Local Fields Potentials
MeSH Terms: conditions — Cluster Headache; Trigeminal Autonomic Cephalalgias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Local Field potential recording — Continuous recording of Local Field potentials in patients implanted with Deep brain stimulation

SUMMARY:
The physiopathology of trigeminal-autonomic cephalalgia, and more particularly of cluster headache (CH) is still partially unknown. Three main structures are involved: the trigeminovascular system, the cephalic afferents of the autonomic nervous system, and centrally the hypothalamus. There are many clinical arguments in favor of the involvement of the hypothalamus in CH. In addition, several radiological studies have confirmed the involvement of the posterior hypothalamic region in cluster attacks. Thus, a positron emission tomography study showed hyperactivity of the posteroinferior nucleus of the ipsilateral hypothalamus. Voxel based MRI studies have shown a bilateral increase in the volume of the inferoposterior part of the homolateral hypothalamus. The involvement of the posterior hypothalamic region or more precisely the ventral tegmental area of the midbrain therefore seems acquired, although its real role as a generator or modulator of pain remains to be precised.

Deep brain stimulation (dBS) is used in the management of chronic drug-resistant CH with an overall efficacy in 2/3 of patients. Nevertheless, its mechanism of action remains poorly understood, thus limiting the selection of patients and the optimization of care. The lack of clear neurophysiological criteria to identify the neuronal population to be targeted is a major source of uncertainty in the positioning of dBS electrodes and parameters adjustment. In order to improve the understanding and at the same time the results of this technique, obtaining in vivo electrophysiological data seems mandatory. Local fields potentials (LFP) have been recordered by in vivo by dBS in other diseases (Parkinson's disease, tremor…) and their analysis has brought new insigights in the characterization and understanding of these pathology. New generations of neurostimulator (Percept Medtronic) enables continuous recording of LFP in implanted patients. The goal of our study is the recording of LFP at the time of CH attacks via the BrainSenseTM system. This system included in the stimulator allows in vivo collection of LFP in the absence and presence of stimulation. The pathophysiological data recordered will then be correlated with the clinical benefit of the dBS ( nulber of attacks, duration, pain intensity…). As it is a feasibility study, only 5 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age : 18-70 years-old) suffering from refractory chronic cluster headache
* Patients eligible for a deep brain stimulation in the ventral tegmental area of the mesencephalon
* Patients implanted with a deep brain stimulation system PerceptTM Medtronic®

Exclusion Criteria:

* Secondary cluster headache
* Patients implanted with another device of deep brain stimulation

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients suffering from refractry chronic cluster headache
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2023-05-31 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Local field potentials | Between 0 to 12 months
  Local field potentials amplitudes registered by the patient during a cluster attack

SECONDARY OUTCOMES:
Change in Efficacy of deep brain stimulation on attacks frequency | Between 0 to 12 months
  Frequency of cluster attacks
Change in Efficacy of deep brain stimulation on pain intensity | Between 0 to 12 months
  Pain intensity of cluster attacks
Change Efficacy of deep brain stimulation in attacks duration | Between 0 to 12 months
  Duration of cluster attacks
Change in Efficacy of deep brain stimulation on treatment | Between 0 to 12 months
  Medical treatments for cluster headache

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided